CLINICAL TRIAL: NCT02949232
Title: Prednisolone Addition for Patients With Recent-onset Psychotic Disorder: the Role of Immune-modulating Strategies in the Treatment of Psychosis
Brief Title: Prednisolone Addition for Patients With Recent-onset Psychotic Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties with recruitment
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Iris Sommer, Prof. Dr., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL46653
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Psychotic Disorder NOS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisolone (Experimental): Prednisolone will be initiated at 40 mg for three days, after which it will be phased out within 6 weeks after start, following treatment guidelines for Inflammatory Bowel Diseases (2008).
  Interventions: Drug: Prednisolone
- Placebo Oral Tablet (Placebo Comparator): Placebo will be initiated at 40 mg for three days, after which it will be phased out within 6 weeks after start, following the treatment schedule of the experimental arm
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Prednisolone — prednisolone will be will be initiated during the first week at 40mg/day for 3 days and 30mg/day for 4 days, followed by a decrease of 5mg/day per week during the remaining 5 weeks; in the second week, patients will use 25 mg/day, in the third week 20 mg/day is used etc. In the last week the patients will only take prednisolone on day 1-3 and day 5 and 7; a tapering scheme in line with the treatment guidelines for Inflammatory Bowel Diseases (2008).
  Arms: Prednisolone
Drug: Placebo Oral Tablet — Dosing following the tapering scheme of the treatment of the treatment arm
  Arms: Placebo Oral Tablet

SUMMARY:
Treatment with prednisolone can be used as a proof of concept to investigate the possibility of immune modulation as a treatment for schizophrenia. It is expected that daily treatment with prednisolone in addition to antipsychotic treatment reduces psychotic symptoms and improves cognition, as compared to placebo. The investigators propose to investigate the effects of administering the corticosteroid prednisolone versus placebo in addition to standard antipsychotic medication in patients with early stage schizophrenia or related disorders, hypothesizing that a decrease in the overall low-grade cerebral inflammation due to prednisolon treatment will be expressed as a decrease in overall symptom severity., Secondly, addition of prednisolone is hypothesised to slow down cognitive deterioration in recent-onset psychosis patients. Finally, the investigators aim to determine whether indirect immunological parameters of the hypothesised low grade inflammation status in schizophrenia are shifted due to the addition of prednisolone.

DETAILED DESCRIPTION:
In the current study, the investigators aim to investigate the effect of additional treatment with prednisolone on symptomatic improvement, global functioning, cognition and on immunological parameters in patients with early-stage psychotic disorder, applying a randomized double-blind placebo-controlled add-on design. A placebo-controlled design was chosen in order to differentiate between clinical effects of prednisolone and effects associated with experimental treatment, such as induced expectations of participants. Prednisolone or placebo is provided next to existent antipsychotic medication as the investigators do not intend to replace existing treatment, this study being a Proof of Concept trial. It would carry considerable risks for patients to taper down existent antipsychotic medication and randomize patients to either placebo or a type of therapy for which the efficacy still has to be proven, even for a short period of time.

90 patients with schizophrenia, schizoaffective or schizophreniform disorder, or psychotic disorder NOS (not otherwise specified) will be included, with an age of 18-70 years and a time interval between the onset of psychosis and study entry not exceeding seven years. All 90 in- and outpatients will be randomized 1:1 to either prednisolone or placebo daily for 6 weeks. Prednisolone will be initiated at 40mg/day for 3 days and the 4 remaining days of the first week 30mg/dag will be used. During the treatment period, patients will be seen at weekly intervals to assess symptom severity, depressive mood and suicidal ideation, global functioning and side effects.

ELIGIBILITY:
Inclusion Criteria:

1. A DSM-IV-R diagnosis of: 295.x (schizophrenia, schizophreniform disorder, or schizoaffective disorder) or 298.9 (psychosis NOS)
2. Onset of psychosis no longer than 7 years ago
3. Minimum total PANSS score of 60
4. Age 18 -70 years
5. Patients are treated with antipsychotic medication
6. Written informed consent is obtained
7. Female patients of childbearing potential need to utilize a proper method of contraception (the pill, vaginal ring, hormonal patch, intrauterine device, cervical cap, condom, contraceptive injection, diaphragm) in case of sexual intercourse during the study.

Exclusion Criteria:

1. Presence of any of the contra-indications of prednisolone as reported in the SPC.
2. Presence of diabetes mellitus or random (non-fasting) glucose levels exceeding 11 mmol/L at screening, severe heart failure, severe osteoporosis or systemic fungal infections.
3. Body Mass Index (BMI) of >30.0
4. Current or chronic use of systemic glucocorticosteroids (temporary use is permitted, if stopped 1 month before start of treatment trial)
5. Chronic use of non-steroidal anti-inflammatory drugs, defined as daily use during more than 2 months. Intermittent use is permitted, if stopped at least 1 month before start of treatment trial.
6. Pregnancy or breast-feeding. A urine pregnancy test will be performed at screening.
7. Concurrent use of certain types of medication:

1. liver enzyme inducing medication such as carbamazepine, riphampicine, primidone, barbiturates and phenytoine

2. HAART medication (both HIV protease inhibitors and (non)-nucleoside reverse transcriptase inhibitors), especially efavirenz, ritonavir and lopinavir.

3. telaprevir and boceprevir in treatment of Hepatitis C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change in symptom severity | 6 weeks
  Change in symptom severity is expressed as a change in total score on the Positive and Negative Symptom Scale (PANSS) from baseline to end of the 6-week treatment.

SECONDARY OUTCOMES:
Improvement in cognitive functioning | 6 months
  Cognitive functioning is measured through the Brief Assessment of Cognition in Schizophrenia (BACS).
Change in GAF scores | 1 year
  Global Assessment of Functioning
Measurement of various immunological biomarkers | 6 months
  Cytokine panels will be analysed
Improvement of PANSS scores in follow-up | 1 year
  PANSS follow-up; 4 months, 6 months and 12 months
Score on the Calgary Depression Scale for Schizophrenia (CDSS) | 6 weeks
  CDSS scores will be analysed
Incidences of key SAEs and SUSARs | 1 year
  Safety analyses

CONTACTS AND LOCATIONS:
Overall Officials: Iris Sommer, Prof. Dr., Principal Investigator — UMC Utrecht
Locations (4):
- ZNA, Antwerp, Belgium
- University Aarhus, Risskov, Denmark
- Netherlands (2):
  - Yulius, Sliedrecht
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nasib LG, Gangadin SS, Rossum IW, Boudewijns ZSRM, de Witte LD, Wilting I, Luykx J, Somers M, Veen N, van Baal C, Kahn RS, Sommer IE. The effect of prednisolone on symptom severity in schizophrenia: A placebo-controlled, randomized controlled trial. Schizophr Res. 2021 Apr;230:79-86. doi: 10.1016/j.schres.2021.01.024. Epub 2021 Mar 10. PMID 33711681